CLINICAL TRIAL: NCT03575689
Title: The Efficacy of Silastic Sheet Nasal Splints in Endoscopic Nasal Septal Repair Surgery: A Prospective Randomized Control Trial
Brief Title: Nasal Splint and Endoscopic Nasal Septal Repair Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Paul's Hospital, Canada (Other)
Responsible Party: Principal Investigator, Amin Javer, Director, St. Paul's Sinus Centre, St. Paul's Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H15-03025
Record Dates: First submitted 2018-06-19; First posted 2018-07-02 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Septum Deviated
Keywords: Nasal Splint; Septum deviation; Septoplasty

STUDY DESIGN:
Intervention Model Description: There will be two possible scenarios resulting from randomization: All patients will undergo septoplasty using quilting technique.
  A. The Doyle splint will be places in both nostrils of the patient after septoplasty. The doyle splints will be removed 6 days after surgery as per standard of care. No other procedures will be changed during the surgery.
  B. No Doyle splints will be placed in the nostrils of the patient after septoplasty. All standart of care visits will remain the same.
Who Masked: Outcomes Assessor
Masking Description: The PI will be the blinded assessor. The choice of which patient gets a Doyle splint will be randomized using the sealed envelope system mentioned above.
  The randomization will be balanced to ensure that both arms have patients with extensive surgeries as well as isolated NSRs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Splint (Experimental): A. The Doyle splint will be places in both nostrils of the patient after septoplasty. The doyle splints will be removed 6 days after surgery as per standard of care. No other procedures will be changed during the surgery.
  Interventions: Device: Doyle Splint
- No Splint (No Intervention): B. No Doyle splints will be placed in the nostrils of the patient after septoplasty. All standart of care visits will remain the same.

INTERVENTIONS:
Device: Doyle Splint — Using Doyle splints following septoplasty is the standard of care and may help with stability of the septum in the immediate post op period. owever these splints are associated with morbidity in the post-op period. The quilting technique was developed to prevent complications and stabilize the septum. This study examines the efficacy of these splints in stabilizing the septum and preventing complications after septoplasty
  Arms: Splint

SUMMARY:
Septoplasty is one of the most performed surgeries in rhinology as a solo procedure, or in combination with sinus surgery. The procedure for septoplasty and postoperative management has evolved over time based on several studies that have been done. The current standard of care in our centre is to conduct a septoplasty using quilting technique and apply Doyle splints in both nostrils to stabilize the septum for 6 days. However these splints are associated with morbidity in the post-op period. The quilting technique was developed to prevent complications and stabilize the septum. This study examines the efficacy of these splints in stabilizing the septum and preventing complications after septoplasty

DETAILED DESCRIPTION:
1. Purpose

   To compare the success rate of septoplasty in correcting the nasal septal deviation (with regards to nasal obstruction and intranasal access) among patient who used Doyle splints and those who did not. The investigators will also determine if patient's quality of life in the postoperative period is affected by the use of Doyle splints or not.
2. Hypothesis

   Is there a significant difference in success rates of septoplasty in patients who used a Doyle nasal splint when compared with patients who did not use the Doyle nasal splint? Null hypothesis There is no significant difference in success rates of septoplasty in patients who used a Doyle nasal splint when compared with patients who did not use the Doyle nasal splint.
3. Justification

   Currently in most North American rhinology clinics, nasal splints are used after septoplasty (using the quilting technique) to improve stability of the nasal septum. The quilting technique in addition to reduction of other complications was developed to improve septal stability after septoplasty. No study has been conducted to examine the efficacy of using only the quilting method when compared to the current standard of care which adds extra cost to the surgery. This study aims to evaluate the efficacy of the quilting technique in improving stability of the nasal septum among patients using nasal splints and those not on nasal splints after septoplasty.

   A recent study (Objective usefulness of thin silastic septal splints after septal surgery; i Jung, M.D., Kim, M.D. et al Am J Rhinol Allergy 25, 182-185, 2011) has shown Insertion of a silastic septal splint after septal surgery should be accepted as a routine procedure. Our study is aiming to show that quilting suture in x-shaped fashion technique is as effective and safe as using them yet avoids the potential complication of discomfort/pain/toxic shock syndrome etc.

   The essence of this study is to show that using the quilting suture technique alone without splints is as good as when used with splints. No other study has been done to investigate this.
4. Objectives

   Primary Objective To compare the success rate of septoplasty in correcting the nasal septal deviation (with regards to nasal obstruction and intranasal access) among patient who used Doyle splints and those who did not.

   Secondary Objectives To determine if patient's quality of life in the postoperative period is affected by the use of Doyle splints or not.
5. Research Method

   This is a Single blind Randomized Control Trial.

   Procedure

   The study population will be consecutive patients diagnosed with nasal septal deviation and who are undergoing nasal septal surgery. It will be a single blind randomized control trial. Allocation concealment will be ensured by the use of sequentially numbered, opaque, sealed envelopes. An assessor blinded to which patient is using Doyle splints will assess the primary outcome.

   Consent will be obtained for this study prior to the surgery.

   Blinding The study will be single-blinded study. The patients will be randomized into 2 arms/groups. An assessor blinded to which patient got the Doyle splints will assess the primary outcome.

   There will be two possible scenarios resulting from randomization: All patients will undergo septoplasty using quilting technique.

   A. The Doyle splint will be places in both nostrils of the patient after septoplasty. The doyle splints will be removed 6 days after surgery as per standard of care. No other procedures will be changed during the surgery.

   B. No Doyle splints will be placed in the nostrils of the patient after septoplasty. All standart of care visits will remain the same.

   The PI will be the blinded assessor. The choice of which patient gets a Doyle splint will be randomized using the sealed envelope system mentioned above.

   The randomization will be balanced to ensure that both arms have patients with extensive surgeries as well as isolated NSRs
6. Statistical Analysis

Sample size calculations Due to lack of data on failure rates of septoplasty in our centre, an a priori sample size calculation was used to determine the number of participants required to adequately compare the use of nasal splints. Given that this clinical trial is designed to investigate equivalency between the use of nasal splints and the lack thereof, an equivalency sample size calculation was performed. An equivalency limit of 5% was considered clinically significant from consultation with our expert rhinologist. A previously conducted study estimating failure and revision rates have estimated that the failure rate was 8%16. If there is truly no difference between the use of splints or lack thereof, then 88 patients (44 patients per group) will be required to be 80% sure that the limits of a two-sided confidence interval will exclude a difference in means of more than 5%. Accounting for dropout rates of 10%, a total of 96 patients (48 patients per group) will be required for this study.

Statistical Comparisons The primary objective of this randomized controlled trial will be to compare the success rates of septoplasty in patents with and without use of nasal splints up to 90 days post-surgery. Count and absolute percentages of rates will be reported. The Chi-Squared test will be used to determine statistical significance between rates. Probability values less than 5% (α=0.05) will be considered significant. Corresponding odds ratios and 95% confidence intervals will be reported.

For the secondary outcome measures (e.g. VAS, NOSE), results will be summated and considered as continuous, numerical variables. Descriptive statistics using mean, median, standard deviation and inter-quartile ranges will be reported. The unpaired two sample student t-tests will be applied to investigate the difference between the means of the various outcome measures. Probability values less than 5% (α =0.05) will also be considered statistically significant.

Baseline demographics and clinical factors will be compared between each treatment group to determine whether randomization yielded comparable groups. Multivariable logistic and linear regression will be used to investigate the relationships in the primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients 19 years and above diagnosed with deviated nasal septum using the Mladina septal deviation scale who are complaining of nasal obstruction and/or sinus disease
* These patients will also be undergoing a nasal septoplasty either as a standalone case or as part of endoscopic sinus surgery and/or resection of the inferior turbinates. These surgeries could either be a primary or revision case.

Exclusion Criteria:

* Patients with sinonasal tumors
* Cystic fibrosis or syndromic patients (e.g. Wegeners granulomatosis, immunocompromised)
* Patients with autoimmune diseases
* Patients who do not understand English language and to understand the purpose, methods and conduct of this study.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2016-03-24 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Mladina | 3 months for every patient
  Mladina Classification of Septal Deformity: This test will be performed by same blinded assessor before and after the surgery. This is a validated and widely used system for classifying nasal septal deviation.

SECONDARY OUTCOMES:
Visual Analog Scale | 3 months for every patient
  Pain and discomfort (Visual Analog Scale): The visual analog score describes subjective pain and discomfort levels experienced by the participant following the procedures in both arms of the study.
  The scoring would be : 0-10 for the subscales and 0-50 for the total pain VAS score; 0 is best 10 is the worst score. Subscales will be summed.
Postoperative complications | 3 months for every patient
  Postoperative complications: The following complications will be evaluated on a present/absent basis.
  * Hemorrhage
  * Hematoma formation
  * Adhesion formation (Between the middle turbinate and nasal septum)
  * Septal Perforation

CONTACTS AND LOCATIONS:
Overall Officials: Amin Javer, MD FRCSCFARS, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - E.N.T. Clinic, St. Paul's Hospital, Vancouver, British Columbia
  - St Paul Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: Undecided